CLINICAL TRIAL: NCT01120821
Title: A Phase II Trial of the Treatment of Polycythemia Vera With Gleevec
Brief Title: Treatment of Polycythemia Vera With Gleevec
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Richard Silver, M.D., Weill Cornell Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702-375; CSTI571AUS41 (Other Grant/Funding Number: Novartis)
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Polycythemia Vera
Keywords: PV
MeSH Terms: conditions — Polycythemia Vera | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study drug (Experimental): Gleevec treatment
  Interventions: Drug: Gleevec

INTERVENTIONS:
Drug: Gleevec — 400 mg once daily for 12 months
  Other Names: STI-571

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of patients with Polycythemia Vera treated with Gleevec.

DETAILED DESCRIPTION:
Phlebotomy is a standard temporizing treatment for Polycythemia Vera. Performing repeated phlebotomies may lead to iron deficiency and can contribute to a rising platelet count. This may create additional problems, such as clots particularly in patients older than 50. There is reason to believe that the use of Gleevec may cause a decrease in the activity of the marrow so that patients may not require as many or any phlebotomies. Thus, spleen function may possibly improve by decreasing in size and patients' platelet counts may also improve.

ELIGIBILITY:
Inclusion Criteria:

* Patients have diagnosis of Polycythemia Vera (PV). Patients may have newly diagnosed PV.
* Patients may have previously interferon-alfa treated PV with documented resistance, refractoriness or intolerance to interferon-alfa.
* Patients may have PV with inadequate control on hydroxyurea.
* Performance status of 0, 1, or 2
* Adequate end organ function, defined as the following:

  1. total bilirubin <1.5 x upper limit of the normal range (ULN)
  2. SGOT (AST) and SGPT (ALT) < 2.5 x ULN
  3. creatinine < 1.5 x ULN
  4. ANC > 1.5 x 109/L
* Written voluntary informed consent.

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding.
* Patients receiving busulfan within 6 weeks of Study Day 1.
* Patients receiving interferon-alpha within 4 weeks of Study Day 1.
* Patients receiving hydroxyurea within 2 weeks of Study Day 1.
* Patients with Grade III or IV cardiac problems as defined by the New York Heart Association Criteria.
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.
* Patients previously treated with Gleevec.
* Serum erythropoietin level > or = 25 units/microliter
* Abnormal O2 saturation (by pulse oximetry) or arterial pO2 (by arterial blood gas).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-08; Primary Completion 2007-01 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Stabilization of hematocrit | Weekly for the first six week of treatment, then monthly for one year from study entry.
Platelet count maintenance a therapeutic range. | Weekly for the first six weeks of treatment, then monthly for one year from study entry.

SECONDARY OUTCOMES:
Splenomegaly (if existent) | Weekly for the first six weeks of treatment, then montly for one year from study entry.
Quality of life, performance status, side effects and complications during treatment. | Weekly for the first six weeks of treatment, then montly for one year from study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Silver, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States